CLINICAL TRIAL: NCT04130360
Title: A Randomized Controlled Trial of an Online Problem-solving Intervention to Reduce Aggression Among Youth
Brief Title: A Trial of an Online Problem-solving Intervention for Aggression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 030755
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2019-10

CONDITIONS: Aggression
Keywords: problem-solving; youth; brief intervention; online intervention; young people; aggressive behaviour
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Intervention Model Description: Intervention and control group. Participants are randomised to one of them.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are not told that they are being randomised or that they are participating in an intervention trial until they complete the follow-up. Randomisation is computerized and participants have no contact with a care provider or an investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem-solving (Experimental)
  Interventions: Behavioral: Problem-solving
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Problem-solving — The steps of problem-solving are explained to the participants. Then, they are presented two conflictive situations and they are asked to apply the problem-solving steps to find a solution. Once they finish, they are asked to apply the steps in a conflictive situation they have experience in the last month. In the end, they are reminded of the steps and encouraged to practice them in their daily conflicts.
  Other Names: social problem-solving
  Arms: Problem-solving

SUMMARY:
Aggressive behaviour among adolescents is a social problem that can be reduced by social problem-solving interventions. However, these interventions usually include more than one technique, and the specific techniques that are effective in reducing and preventing aggression remain to be identified. Therefore, the main aim of this study is to test whether the instruction and practice of problem-solving on their own are effective in changing aggressive behaviour among adolescents.

As the intervention in this trial is aimed at the general population, it will be delivered online. The rapid growth in the use of the Internet among young people provides an opportunity to deliver interventions universally in a cheap and efficient way.

Problem-solving skills are fundamental to effective behaviour change. Therefore, problem-solving skills will be measured to assess whether they mediate the effect of the intervention on aggressive behaviour.

Finally, young people with callous-unemotional traits are less likely to change their problematic behaviour such as aggression after an intervention. Therefore, Callous-Unemotional traits will be measured to assess if they act as a moderator of effectiveness.

It is expected that participants randomised to the intervention improve their problem-solving skills and consequentially, reduce their aggressive behaviours. In addition, participants with lower callous-unemotional traits are expected to have a greater change.

ELIGIBILITY:
Inclusion Criteria:

* Living in the UK
* Fluent in English

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 908 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Aggression (trait) | 1 month
  Aggression Questionnaire (AQ): Physical Aggression, Verbal Aggression, Hostility, Anger. Each item is responded from 1 (extrememly uncharacteristic of me) to 5 (extremely characteristic of me), with higher scores meaning higher aggression.
Aggression (frequency) | 1 month
  Physical and relational aggression questionnaire. Each item is responded from 1 (never) to 5 (5 or more times), with higher scores meaning higher aggression.

SECONDARY OUTCOMES:
Problem-solving skills | 1 month
  Problem Solving Skills (PSI-PSS). Each item is responded from 1 (strongly disagree) to 6 (strongly agree), with higher scores meaning higher problem-solving skills.
Problem-solving self-efficacy | 1 month
  Problem Solving Self-Efficacy (PSI-PSSE). Each item is responded from 1 (strongly disagree) to 6 (strongly agree), with higher scores meaning higher problem-solving self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Castillo-Eito, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data will be shared, but there is not a concrete plan at the moment.